CLINICAL TRIAL: NCT04673643
Title: Transcutaneous Auricular Vagus Nerve Stimulation in Dry Eye Disease: A Randomized Clinical Trial
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation in Dry Eye Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, wudong0120, Doctor, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: taVNS-DED-2020
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dry Eye Disease
Keywords: taVNS; Dry eye; RCT
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Transcutaneous Auricular Vagus Nerve Stimulation
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS group (Experimental): taVNS device (Elmmedicare, EC100, Shenzhen, China) was used to apply stimulation for patients. Stimulation parameters comprised an electrical current of 1 mA at a frequency of 20 Hz, with a waveform width of 1 ms. Repurposed off-the-shelf devices were utilized for this purpose, with the stimulator generating single square-wave pulses lasting 1 ms each. Enhancing conductivity was achieved by wiping the ear with tap water. The electrodes were placed on the cymba conchae and concha around the affected ear, which is the region of rich vagus nerve branch distribution.
  Drug: Hyaluronic acid eye drops Participants in both groups received hyaluronic acid eye drops (HYLO COMOD® eye drops, Ursapharm, Ltd., Germany) with the treatment of 3 times a day.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation; Drug: Hyaluronic acid eye drops
- Control Group (Placebo Comparator): taVNS device were applied using the same stimulator, stimulation parameters and same sessions. However, the electrodes were placed on the antihelix around the affected ear, which is the region of few vagus nerve branch distribution. Drug: Hyaluronic acid eye drops Participants in both groups received hyaluronic acid eye drops (HYLO COMOD® eye drops, Ursapharm, Ltd., Germany) with the treatment of 3 times a day.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation; Drug: Hyaluronic acid eye drops

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — taVNS device (Elmmedicare, EC100, Shenzhen, China) was used to apply stimulation for patients.
  Stimulation parameters comprised an electrical current of 1 mA at a frequency of 20 Hz, with a waveform width of 1 ms. Repurposed off-the-shelf devices were utilized for this purpose, with the stimulator generating single square-wave pulses lasting 1 ms each. Enhancing conductivity was achieved by wiping the ear with tap water. The electrodes were placed on the cymba conchae and concha around the affected ear, which is the region of rich vagus nerve branch distribution. Patients in control group were applied using the same stimulator, stimulation parameters and same sessions. However, the electrodes were placed on the antihelix around the affected ear, which is the region of few vagus nerve branch distribution.
Drug: Hyaluronic acid eye drops — Participants in both groups received hyaluronic acid eye drops (HYLO COMOD® eye drops, Ursapharm, Ltd., Germany) with the treatment of 3 times a day.

SUMMARY:
Objective: To evaluate the effect of transcutaneous auricular vagus nerve stimulation (taVNS) for the patients with dry eye disease with meibomian gland dysfunction.

Methods: We enrolled 256 patients at Beijing Tongren Hospital. Patients completed questionnaires at baseline, 1 month, 3 months, and 6 months.OSDI score, TBUT, Schirmer I, tCFS, MGD score, and psychological status to evaluate the therapeutic effects. A difference of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 and Age <=75.
2. Clinical diagnosis of dry eye disease.

Exclusion Criteria:

1. History of depression, tumors, thyroid disease, diabetes, cardiac diseases.
2. History of phthalmology surgery.
3. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
OSDI | Baseline, month 1, 3, and 6
  Ocular Surface Disease Index (OSDI) questionnaire: The OSDI questionnaire is designed to assess the severity of symptoms and the impact of ocular surface diseases, such as dry eye disease, on a patient's quality of life.

SECONDARY OUTCOMES:
TBUT | Baseline, month 1, 3, and 6
  Tear Breakup Time (TBUT): TBUT is a diagnostic test used to evaluate the stability of the tear film and diagnose dry eye disease. It measures the time it takes for dry spots to appear on the corneal surface after blinking while using a fluorescent dye. A shorter TBUT indicates less stable tear film, which is often associated with dry eye disease.
Schirmerl | Baseline, month 1, 3, and 6
  The Schirmer I test assesses tear production to diagnose dry eye syndrome. The length of the wetting is measured in millimeters. A lower measurement indicates reduced tear production, suggesting dry eye disease.
Corneal fluorescein staining (tCFS) | Baseline, month 1, 3, and 6
  tCFS used to assess the damage to the corneal epithelium, particularly in cases of dry eye disease, ocular surface disorders, or trauma.
Meibomian Gland Dysfunction Score | Baseline, month 1, 3, and 6
  MGD score used to assess the function of the Meibomian glands and the overall health of the eyelid margins.
Psychological status | Baseline, month 3, 6 and 12
  9-item Patient Health Questionnaire and Symptom Checklist-90 for anxiety are used to assess the psychological status.

CONTACTS AND LOCATIONS:
Overall Officials: Haihong Lian, Doc, Principal Investigator — BeijingTongren Hospital, Capital Medical University
Locations (2):
- China (2):
  - Beijing Tongren Hospital, Beijing
  - Wu Dong, Beijing